CLINICAL TRIAL: NCT05263505
Title: Baricitinib for the Treatment of Ocular Mucous Membrane Pemphigoid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Michael Paley, Instructor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202107009
Record Dates: First submitted 2022-02-16; First posted 2022-03-02 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Mucous Membrane Pemphigoid; Cicatrizing Conjunctivitis
MeSH Terms: conditions — Pemphigoid, Benign Mucous Membrane | interventions — baricitinib; Methotrexate; Azathioprine; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): 4mg daily
  Interventions: Drug: Baricitinib 2 MG [Olumiant]
- Antiproliferative (Active Comparator): methotrexate, azathioprine, or mycophenolate
  Interventions: Drug: Methotrexate; Drug: Azathioprine; Drug: Mycophenolate

INTERVENTIONS:
Drug: Baricitinib 2 MG [Olumiant] — Two tabs daily
  Arms: Baricitinib
Drug: Methotrexate — Target dose: 20mg weekly
  Arms: Antiproliferative
Drug: Azathioprine — Target dose: 2mg/kg daily
  Arms: Antiproliferative
Drug: Mycophenolate — Target Dose: 1g twice daily
  Arms: Antiproliferative

SUMMARY:
Ocular mucous membrane pemphigoid (MMP) is an autoimmune, scarring conjunctivitis that can lead to vision loss and permanent disability. It is a rare disorder with an estimated incidence of 1 in 60,000. There are currently no FDA-approved medications for the treatment of mucous membrane pemphigoid, highlighting a clear unmet need.

At present, moderate to severe disease requires off-label use of potent immunosuppressive agents, such as oral anti-proliferatives (methotrexate, azathioprine, and mycophenolate), rituximab (RTX) or cyclophosphamide (CyC). Recently, Janus kinase (JAK) inhibition with baricitinib or tofacitinib been reported to be successful in one case of ocular MMP.

This is a randomized, single-masked, two-arm study of baricitinib vs anti-proliferatives for ocular MMP.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet all the following criteria:

Type of Patient and Disease Characteristics

1. Are at least 18 years of age
2. Have a clinical diagnosis of Ocular Mucous Membrane Pemphigoid

   a. The treating ophthalmologist will have excluded alternative etiologies that can cause cicatrizing conjunctivitis such as:
   * Rosacea
   * Atopic dermatitis
   * Lichen Planus
   * Iatrogenic interventions, e.g. glaucoma eye drops
   * Stevens-Johnsons Syndrome
   * Graft vs Host Disease
3. Have active disease based on ophthalmologic exam

   Patient Characteristics
4. Nonpregnant, nonbreastfeeding female or male patient

   1. Female patients of child-bearing potential who are abstinent (if this is complete abstinence, as their preferred and usual lifestyle) or in a same-sex relationship (as part of their preferred and usual lifestyle) must agree to either remain abstinent or stay in a same-sex relationship without sexual relationships with the opposite sex.
   2. Total abstinence is defined as refraining from intercourse during the entirety of the study and for at least 1 week following the last dose of investigational product. Periodic abstinence such as calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception.
   3. Otherwise, female patients of childbearing potential must agree to use 2 effective methods of contraception, where at least 1 form is highly effective, for the entirety of the study and for at least 1 week following the last dose of investigational product.
   4. The following contraception methods are considered acceptable (the patient should choose 2, and 1 must be highly effective [defined as less than 1% failure rate per year when used consistently and correctly]):

      * Highly effective birth control methods:

        * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
        * Progestogen- only containing hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
        * intrauterine device (IUD)/intrauterine hormone-releasing system (IUS)
        * vasectomized male (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
      * Effective birth control methods:

        o Male or female condom with spermicide. It should be noted that the use of male and female condoms as a double barrier method is not considered acceptable due to the high failure rate when these methods are combined.
      * Diaphragm with spermicide
      * Cervical sponge
      * Cervical cap with spermicide Note: When local guidelines concerning highly effective or effective methods of birth control differ from the above, the local guidelines must be followed.

   Female patients of non-child-bearing potential are not required to use birth control and they are defined as:
   * Women who are infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation)
   * Post-menopausal - defined either as

     o A woman at least 50 years of age with an intact uterus, not on hormone therapy, who has either
   * Cessation of menses for at least 1 year
   * At least 6 months of spontaneous menorrhea with follicle-stimulating hormone >40 mIU/mL

     * Women aged 55 years or older who are not on hormone therapy, and who have had at least 6 months of spontaneous amenorrhea
     * Women aged 55 years or older who have a diagnosis of menopause

   Informed Consent
5. Must read and understand the informed consent approved by the institutional review board (IRB)/ethics review board (ERB) governing the site and provide written informed consent.

   Exclusion Criteria:

   Patients will be excluded from study enrollment if they meet any of the following criteria:

   Disease Characteristics
6. Have rapidly progressive disease, as determined by the treating ophthalmologist, that places the patient at an unacceptable risk for participating in the study

   Medical Conditions
7. Have had any major surgery within 8 weeks prior to screening or will require major surgery during the study that, in the opinion of the investigator would pose an unacceptable risk to the patient.
8. Have experienced any of the following within 12 weeks of screening: VTE (DVT/pulmonary embolism [PE]), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
9. Have a history of recurrent (≥ 2) VTE (DVT/PE).
10. Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
11. Have a history of lymphoproliferative disease; have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years prior to randomization.

    The following may be exempted:
    1. Patients with cervical carcinoma in situ that has been resected with no evidence of recurrence or metastatic disease for at least 3 years may participate in the study.
    2. Patients with basal cell or squamous epithelial skin cancers that have been completely resected with no evidence of recurrence for at least 3 years may participate in the study.
12. Have a current or recent (<4 weeks prior to randomization) clinically serious viral, bacterial, fungal, or parasitic infection or any other active or recent infection that in the opinion of the investigator, would pose an unacceptable risk to the patient if participating in the study.

    Note: For example, a recent viral upper respiratory tract infection or uncomplicated urinary tract infection need not be considered clinically serious.
13. Have symptomatic herpes simplex at the time of randomization
14. Have had symptomatic herpes zoster infection within 12 weeks prior to randomization
15. Have a history of disseminated/complicated herpes zoster (for example, ophthalmic zoster or CNS involvement).
16. Have a positive test for hepatitis B virus (HBV) defined as:

    1. positive for hepatitis B surface antigen (HBsAg), or
    2. positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA)

    Note: Patients who are HBcAb-positive and HBV DNA-negative may be enrolled in the study but will require additional HBV DNA monitoring during the study.
17. Have hepatitis C virus (HCV) infection (hepatitis C antibody-positive and HCV ribonucleic acid [RNA]-positive).

    Note: Patients who have documented anti-HCV treatment for a past HCV infection AND are HCV RNA-negative may be enrolled in the study.
18. Have evidence of HIV infection and/or positive HIV antibodies
19. Have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB
20. Have evidence of active TB or latent TB

    1. Have evidence of active TB, defined in this study as the following:

       * Positive purified protein derivative (PPD) test (≥5 mm induration between approximately 2 and 3 days after application, regardless of vaccination history), medical history, clinical features, and abnormal chest x-ray at screening
       * QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. Patients are excluded from the study if the test is not negative and there is clinical evidence of active TB

       Exception: patients with a history of active TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, have no clinical features of active TB, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT®.TB test but must have a chest x-ray at screening (i.e., chest imaging performed within the past 6 months will not be accepted).
    2. Have evidence of untreated/inadequately or inappropriately treated latent TB, defined in this study as the following:

       * Positive PPD test, no clinical features consistent with active TB, and a chest x-ray with no evidence of active TB at screening; or
       * If the PPD test is positive and the patient has no medical history or chest x-ray findings consistent with active TB, the patient may have a QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines). If the test results are not negative, the patient will be considered to have latent TB (for purposes of this study); or
       * QuantiFERON®-TB Gold test or T- SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. If the test results are positive, the patient will be considered to have latent TB. If the test is not negative, the test may be repeated once within approximately 2 weeks of the initial value. If the repeat test results are again not negative, the patient will be considered to have latent TB (for purposes of this study).

    Exception: Patients who have evidence of latent TB may be enrolled if he or she completes at least 4 weeks of appropriate treatment prior to randomization and agrees to complete the remainder of treatment while in the trial.

    Exception: Patients with a history of latent TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, have no clinical features of active TB, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT®.TB test but must have a chest x-ray at screening (i.e., chest imaging performed within the past 6 months will not be accepted).
21. Have received any of the following medications:

    1. Cyclophosphamide (or any other cytotoxic agent) within 4 weeks of screening.
    2. Rituximab or any other B cell depleting therapies within 12 weeks of screening.
22. Have been treated with probenecid that cannot be discontinued for the duration of the study.
23. Have been exposed to a live vaccine within 12 weeks of randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination).

    Note: All patients who have not previously received the herpes zoster vaccine by screening will be encouraged (per local guidelines) to do so prior to randomization; vaccination with live herpes zoster vaccine must occur >4 weeks prior to randomization and start of investigational product. Patients will not be randomized if they were exposed to a live herpes zoster vaccination within 4 weeks of planned randomization. Investigators should review the vaccination status of their patients and follow the local guidelines for vaccination of patients ≥18 years of age with nonlive vaccines intended to prevent infectious disease prior to entering patients into the study.
24. Are currently enrolled in or have discontinued within 4 weeks of screening from any other clinical trial involving an investigational product or nonapproved use of a drug or device or any other type of medical research judged not to be scientifically or medically compatible with this study.
25. Have screening laboratory test values, including thyroid-stimulating hormone (TSH), outside the reference range for the population that, in the opinion of the investigator, pose an unacceptable risk for the patient's participation in the study. Patients who are receiving thyroxine as replacement therapy may participate in the study, provided stable therapy has been administered for ≥12 weeks and TSH is within the laboratory's reference range. Patients who have TSH marginally outside the laboratory's normal reference range and are receiving stable thyroxine replacement therapy may participate if the treating physician has documented that the thyroxine replacement therapy is adequate for the patient
26. Have any of the following specific abnormalities on screening laboratory tests from the central or local laboratory

    1. ALT or AST >2 x upper limits of normal (ULN)
    2. alkaline phosphatase (ALP) ≥2 x ULN
    3. total bilirubin ≥1.5 x ULN
    4. hemoglobin <10 g/dL (100.0 g/L)
    5. total white blood cell count <3000 cells/μL (<3.00 x 103/μL or <3.00 billion/L)
    6. neutropenia (absolute neutrophil count [ANC] <1500 cells/uL) (<1.50 x 103/uL or <1.50 billion/L)
    7. lymphopenia (lymphocyte count <1000 cells/uL) (<1.00 x 103/μL or <1.00 bilion/L)
    8. thrombocytopenia (platelets <100,000 cells/uL) (<100 x 103/μL or <100 billion/L)
    9. eGFR <60 mL/min/1.73 m2 (Bedside Schwartz formula 2009) In the case of any of the aforementioned laboratory abnormalities, the tests may be repeated once during screening, and values resulting from repeat testing may be accepted for enrollment eligibility if they meet the eligibility criterion

    Other Exclusions
27. Are largely or wholly incapacitated permitting little or no self-care, such as being bedridden or confined to wheelchair
28. In the opinion of the investigator, are at an unacceptable risk for participating in the study
29. Have donated more than a single unit of blood within 4 weeks prior to screening or intend to donate blood during the course of the study
30. Have a history of intravenous drug abuse, other illicit drug abuse, or chronic alcohol abuse within the 2 years prior to screening or are concurrently using, or expected to use during the study, illicit drugs (including marijuana)

    Note: Patients who are prescribed medical marijuana by a physician are not excluded from the study.
31. Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures
32. Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital / Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baricitinib | Antiproliferative
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baricitinib | Antiproliferative | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: Treatment response of ocular inflammation based on conjunctival injection measured by ophthalmologic exam of the palpebral conjunctiva. Each eye is divided into quadrants and each quadrant is scored from 0 (white and quite) to 3 (severe). The score will be the sum of all 4 quadrants for a total score of 0-12 for each eye. A clinically meaningful response will be defined as a ≥30% reduction in the total score for both eyes.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Baricitinib | Antiproliferative
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Averse events were recorded for 2 weeks for the participant in the standard of care arm and 8 months for the participant on the baricitinib arm.
Arm/Group | Baricitinib | Antiproliferative
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (N=1) | Antiproliferative (N=1)
Anaphylaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Prostate Cancer

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT05263505/Prot_SAP_000.pdf